CLINICAL TRIAL: NCT04120766
Title: Safety and Modulation of ABCC9 Pathways by Nicorandil for the Treatment of Hippocampal Sclerosis of Aging: SMArT-HS
Brief Title: Safety and Modulation of ABCC9 Pathways by Nicorandil for the Treatment of Hippocampal Sclerosis of Aging
Acronym: SMArT-HS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gregory Jicha, MD, PhD (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Gregory Jicha, MD, PhD, MD-PhD Professor of Neurology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIA 1R01AG061111; 1R01AG061111 (NIH)
Record Dates: First submitted 2019-10-06; First posted 2019-10-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: TDP-43; Hippocampal sclerosis
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Hippocampal Sclerosis | interventions — Nicorandil

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled, randomized 1:1, single center study of nicorandil (20 mg by mouth daily) or placebo for 96 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled, randomized 1:1, single center study of nicorandil (20 mg by mouth daily) or placebo for 96 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Nicorandil 20mg qd
  Interventions: Drug: Nicorandil
- Placebo (Placebo Comparator): Matched placebo qd
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicorandil — 20 mg po qd
  Arms: Treatment
Drug: Placebo — Matching tablet
  Arms: Placebo

SUMMARY:
Widespread recognition of the current and projected impact of the dementia epidemic has spurred research into novel drug discovery efforts. It is well recognized by most that Alzheimer's disease is not the only form of dementia and that beginning to turn attention to other disease states is critically important in order to alleviate this burden on the elderly population today This proposal seeks to further progress in this area through the repurposing an existing drug therapy as a potential treatment for Hippocampal Sclerosis of Aging. This disease is seldom recognized clinically and yet is the number one Alzheimer's disease mimic the confounds are diagnostic and treatment of subjects suffering from dementia and as of yet has no potential therapeutic interventions identified. As such, the proposed study represents a cutting-edge, data-driven, low-cost, exploration of a novel disease relevant pathway that may hold promise for global efforts targeting late life dementia which is a major health priority in America today.

DETAILED DESCRIPTION:
The proposed project is a pilot clinical trial investigating a potential treatment for hippocampal sclerosis of aging (HS-Aging), a prevalent, high-morbidity mimic of Alzheimer's disease (AD). "AD mimics" (diseases with pathologies other than AD but with similar symptoms) are increasingly appreciated to be important causes of dementia. HS-Aging is a major subtype of dementia, affecting ~10-25% of all persons beyond age 85 and is generally misdiagnosed as AD. The primary aims of this study are to test the safety and efficacy of nicorandil for HS-Aging, based on much prior work elucidating a pharmacologically targetable mechanism for this common cause of cognitive decline and dementia in the aging population. Nicorandil is a vasorelaxant drug, used clinically to treat angina and heart disease disease in the elderly, that has not been tested in humans for the prevention or treatment of dementia. The proposed pilot clinical trial represents the first attempt to expedite drug discovery in HS-Aging, and will guide the rational design of future large-scale Phase II & III prevention trials for this prevalent disease that is a major contributor to the personal suffering of patients and caregivers as well as a major cost to health care expenditures in America today. The potential success of this trial will not only help millions within immediately available treatment for their condition but may also ameliorate the booming economic burden of healthcare costs in America today related to late life dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least age 75 years
2. UPDRS ≤ 7
3. Hachinski Ischemic Score ≤ 4
4. CSF profile of "A-T-N+" defined as Aβ(1-42)>250pg/ml; Total Tau>50pg/ml; Phospho-tau<30pg/ml within 24 months, Aβ PET scan negative for Alzheimer's disease within 24 months, or plasma profile of Phospho-tau181 negative for Alzheimer's disease ; hippocampal volume ≤ 1 s.d. below age and gender adjusted mean. Plasma ptau181 levels below 3.0 pg/ml.
5. English-speaking, to ensure compliance with cognitive testing and study visit procedures
6. Involvement of a study partner to supervise medications and compliance with study visits/procedure
7. Stable medical conditions for three months prior to screening visit, with no clinically significant abnormalities of hepatic, renal, and hematologic function defined in the opinion of the investigator
8. Stable medications for 4 weeks prior to screening visit
9. Ability to ingest oral medications
10. Physically acceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests.

Exclusion Criteria:

1. Significant neurologic disease such as Parkinson's disease, stroke, brain tumor, multiple sclerosis or seizure disorder
2. Major depression in past 12 months (DSM-IV criteria)
3. Recent (in past 12 months) substance abuse
4. History of cancer within the past two years, with the exception of non-metastatic prostate or non-melanoma skin cancers such as squamous cell and basal cell carcinomas
5. Contra-indications to lumbar puncture (bleeding disorder, platelet count < 100,000, anticoagulant treatment, major abnormality of the spine that would make LP technically difficult) will exclude the participant from engaging in this optional procedure, but the participant may still participate in the main study using plasma p-tau181 and/or amyloid-PET for Alzheimer's disease screening
6. Use of any investigational agents within 30 days prior to screening
7. Major surgery within eight weeks prior to the Baseline Visit
8. Severe unstable medical illnesses, including uncontrolled cardiac conditions or heart failure (New York Heart Association Class III or IV)
9. Blindness, deafness, or any other disability which may prevent the participant from participating or cooperating in the protocol.

Excluded Medications*

Participants are not eligible for participation in the study if they are taking:

1. Experimental drugs
2. Vasoactive nitrates such as isosorbide dinitrate
3. Drugs for erectile dysfunction such as sildenafil, vardenafil, and tadalafil among others
4. Sulfonylurea antidiabetic agents that may confound efficacy measures for the secondary efficacy outcome measures.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of subjects by arm that experience treatment-related adverse events at week 96 | 96 weeks
  Safety

SECONDARY OUTCOMES:
Hippocampal volume (CC) | 96 weeks
  Change in hippocampal volume over time using freesurfer analyses

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Jicha, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared to other researchers upon request and approval by the study leaders to ensure that data requests do not impinge on the reporting of the primary outcomes or influence study conduct or post conduct analyses. Such IPD will be made available one year following publication of the primary manuscript
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: one year following publishing the primary study results